CLINICAL TRIAL: NCT02475031
Title: Randomized, Prospective, Double Blind Study Comparing Single Shot Versus Continuous Transverses Abdominis Plane (TAP) Block for Postoperative Analgesia After Laparoscopic Live Donor Nephrectomy
Brief Title: Single-shot TAP Block vs Continuous TAP Block
Acronym: TAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Halyard Health (Industry)
Responsible Party: Principal Investigator, Yar Yeap, Assistant Professor of Clinical Anesthesia, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1201007846
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
Keywords: transversus abdominis plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Group (TAP-S) (Placebo Comparator): (TAP-S) - the On-Q reservoir will be filled with saline and set to infuse at rate of 10 ml/hr through the TAP catheter
  Interventions: Drug: TAP-S
- Active Group (TAP-C) (Active Comparator): (TAP-C) - The On-Q reservoir will be filled with 0.2% ropivacaine and set to infuse at rate of 10 ml/hr through the TAP catheter
  Interventions: Device: TAP-C

INTERVENTIONS:
Device: TAP-C — TAP catheters with ropivacaine infusion are inserted into the TAP area after a single shot TAP block. Single shot TAP block is performed using 30ml 0.5% ropivacaine at the end of the case.
  Other Names: Continuous TAP catheter
  Arms: Active Group (TAP-C)
Drug: TAP-S — Catheters with saline infusion are inserted into the TAP area after a single shot TAP block. Single shot TAP block is performed using 30ml 0.5% ropivacaine at the end of the case.
  Other Names: Single shot TAP block
  Arms: Placebo Group (TAP-S)

SUMMARY:
The purpose of this study is to determine whether continuous transversus abdominis plane (TAP) block is superior to single shot TAP for postoperative pain after laparoscopic donor nephrectomy

DETAILED DESCRIPTION:
This study is a randomized, prospective, double blind study comparing single shot versus continuous transversus abdominis plane (TAP) block for postoperative analgesia after laparoscopic live donor nephrectomy.

Good pain control after surgery has been shown to decrease complications. To address the problem of postoperative pain control in donor nephrectomy patients,the study investigators began performing Transversus Abdominis Plane (TAP) blocks. The TAP block involves injection of local anesthetic between the abdominal muscle planes (internal oblique muscle and transversus abdominis muscle), to block the somatic nerves that supply sensation to the skin, muscles, and parietal peritoneum of the anterior abdominal wall. Prior reports of TAP blocks have shown that it provides good analgesia for postoperative pain after abdominal surgery. However because the duration of postoperative pain exceeds that of the single shot TAP block, the investigators hypothesized that by placing a catheter through which a continuous infusion of local anesthetic could be delivered, investigators could provide analgesia throughout the postoperative period. The study investigators also hypothesized that improved analgesia would decrease the need for opioid pain medications, hence decreasing the side effects associated with opioid use.

This study is designed to test our hypothesis that placing a TAP catheter is superior to single shot TAP, because it provides a longer duration of analgesia and decreases narcotic use.

ELIGIBILITY:
Inclusion criteria:

* Healthy subject undergoing laparoscopic live donor nephrectomy
* (ASA) American Society of Anesthesiologists class 1 or 2
* Age 18 or older, male or female
* Desires TAP block for postoperative pain control

Exclusion criteria:

* Any contraindication for TAP block - single or continuous
* History of substance abuse
* Any physical, mental or medical conditions which, in the opinion of the investigators, may confound quantifying postoperative pain resulting from surgery.
* Known allergy or other contraindications to the study medications (Ropivacaine, Normal Saline, Hydromorphone, Oxycodone and Acetaminophen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yar Yeap, MD, Principal Investigator — Indiana University Hospital
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Result] Yeap YL, Wolfe JW, Kroepfl E, Fridell J, Powelson JA. Transversus abdominis plane (TAP) block for laparoscopic live donor nephrectomy: Continuous catheter infusion provides no additional analgesic benefit over single-injection ropivacaine. Clin Transplant. 2020 Jun;34(6):e13861. doi: 10.1111/ctr.13861. Epub 2020 Apr 9. PMID 32198963

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group (TAP-S): (TAP-S) - the On-Q reservoir will be filled with saline and set to infuse at rate of 10 ml/hr through the TAP catheter
  TAP Catheters: Both groups will have catheters inserted into the TAP area after a single shot TAP block
  Placebo: Placebo Group (TAP-S) (TAP-S) - the On-Q reservoir will be filled with saline and set to infuse at rate of 10 ml/hr through the TAP catheter Both groups will receive single shot TAP block with 30ml 0.5% ropivacaine at the end of case
  ropivacaine: The On-Q reservoir will be filled with 0.2% ropivacaine and set to infuse at rate of 10 ml/hr through the TAP catheter Both groups will receive single shot TAP block with 30ml 0.5% ropivacaine at the end of case
  Oxycodone/Acetaminophen
- Active Group (TAP-C): (TAP-C) - The On-Q reservoir will be filled with 0.2% ropivacaine and set to infuse at rate of 10 ml/hr through the TAP catheter
  TAP Catheters: Both groups will have catheters inserted into the TAP area after a single shot TAP block
  ropivacaine: The On-Q reservoir will be filled with 0.2% ropivacaine and set to infuse at rate of 10 ml/hr through the TAP catheter Both groups will receive single shot TAP block with 30ml 0.5% ropivacaine at the end of case
  Oxycodone/Acetaminophen
Period: Overall Study
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C)
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.26 (12.07) | 39.91 (10.21) | 41.09 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 10 | 12 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Total Narcotic Usage at 48 Hours
Description: The primary endpoint of this study will be narcotic requirement at 48 hours
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: mg
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C)
Number analyzed (Participants) | 35 | 35
mg | 2.44 (0.43) | 2.88 (0.59)

2. Secondary Outcome: Secondary Endpoints Measured Will be Total Narcotic Usage at 60 Hours
Description: All narcotic usage will be recorded at 1,12,24,36,48, and 60 hours. All narcotics will be converted to morphine equivalent for statistical calculation. These values reflect the total amount of narcotic used after combining all the data collected from each time point.
Time Frame: up to 60 hours
Measure: Mean (Standard Error); unit: mg
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C)
Number analyzed (Participants) | 35 | 35
mg | 14.31 (2.12) | 14.40 (1.73)

3. Secondary Outcome: Average Pain Scores
Description: Post- operative VAS pain scores (range of 0-10. 0 being no pain and 10 being worst pain) will be recorded at 1,12, 24, 36,48 and 60 hours. The values at each time points were combined and averaged.
Time Frame: up to 60 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C)
Number analyzed (Participants) | 35 | 35
units on a scale | 5.31 (0.34) | 5.06 (0.31)

4. Secondary Outcome: Nausea Scores at 48 Hours
Description: Post-operative nausea scores will be recorded at 48 hours. Range of nausea score is 0-3. 0= None, 1=Mild, 2=Moderate, 3=Severe.
Time Frame: up to 48 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C)
Number analyzed (Participants) | 35 | 35
units on a scale | 0.34 (0.12) | 0.34 (0.11)

5. Secondary Outcome: Sedation Scores at 48 Hours
Description: Post-operative sedation scores will be recorded at 48 hours. Range of score is 0-3. 0=Awake and Alert, 1=Quietly Awake, 2=Asleep and Arousable, 3=Deep sleep.
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C)
Number analyzed (Participants) | 35 | 35
units on a scale | 0.2 (0.08) | 0.06 (0.04)

ADVERSE EVENTS:
Description: Serious and other adverse events were not monitored/addressed.
Arm/Group | Placebo Group (TAP-S) | Active Group (TAP-C)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No